CLINICAL TRIAL: NCT00745680
Title: Morphodynamic Study of Left Ventricular Remodeling With Possible Mechanisms for Pharmacologic Therapy: Assessment by Real-time 3-dimensional Echocardiography and 2-dimensional Speck Tracking Imaging.
Brief Title: Speckle Tracking Imaging and Realtime 3 Dimensional Echocardiograhy to Study LV Function and Remodeling After Acute Myocardial Infarction (AMI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Lung-Chun Lin, National Taiwan University Hospital
Other Study IDs: 200701057R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Congestive Heart Failure; Mitral Regurgitation
Keywords: Left ventricular remodeling, acute myocardial infarction
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: A: AMI patient

SUMMARY:
Left ventricular (LV) remodeling after acute myocardial infarction (AMI) has been well described in previous studies. However, there is a paucity of data on the incidence of and risk factors for LV remodeling in modern clinical practice that incorporates widespread use of acute reperfusion strategies and almost systematic use of "antiremodeling" medications, such as angiotensin-converting enzyme inhibitors and beta blockers. The recent improvements in AMI management do not abolish LV remodeling, which remains a relatively frequent event after an initial anterior wall AMI. As a leading cause of heart failure, postinfarction LV remodeling represents an important target for therapeutic interventions. Within the ventricular mass, size, shape, connections and orientation in a three-dimensional space of every single constituent determine its functional behavior. The complex architecture of the ventricular mass creates multiple inhomogeneities of electrical and mechanical loads at the cellular and the microscopic tissue level, that cause cardiac function to be 'stochastic in nature'. The myocardial infarction will altered the ventricular shape and functional inhomogeneities carrying the morphodynamic advantages such as impaired suction for diastole after diminishing recoil relaxation with decreased twisting strain in systole. The alteration in contractile mechanics interacts with the intraventricular fluid dynamic filed that influence the regional myocardial shearing stress. Altered LV transmural wall strains have been proposed to cause infarct extension and may have an important role in propagating LV remodeling.

DETAILED DESCRIPTION:
We are currently witnessing the advent of new diagnostic tools and therapies for heart diseases, but,without serious scientific consensus on fundamental questions about normal and diseased heart structure and function. During the last decade, three successive, international, multidisciplinary symposia were organized in order to setup fundamental research principles, which would allow us to make a significant step forward in understanding heart structure and function. (Kocica MJ et al., 2006) Helical ventricular myocardial band (HVMB, Figure 2-1) of Torrent-Guasp is the revolutionary new concept in understanding global, three-dimensional, functional architecture of the ventricular myocardium. This concept defines the principal, cumulative vectors, integrating the tissue architecture (i.e. form) and net forces developed (i.e. function) within the ventricular mass. Helical ventricular myocardial band of Torrent-Guasp may also, hopefully, allow overcoming some difficulties encountered in contemporary efforts to create a comprehensive mathematical model of the heart.

Within the ventricular mass, size, shape, connections and orientation in a three-dimensional space of every single constituent determine its functional behavior. This kind of spatial dependence allows the ventricular myocardial mass to be considered as the source of interdependent vectorial forces (i.e.

electrical and mechanical), being generated on different length and time scales. The ultimate net result of these vectorial forces is to translate uniaxial sarcomere shortening into efficient three-dimensional deformation of the ventricular cavity. The complex architecture of the ventricular mass creates multiple inhomogeneities of electrical and mechanical loads at the cellular and the microscopic tissue level, that cause cardiac function to be 'stochastic in nature'. However, at macroscopic (i.e. organ) level, these stochastic events become average and appear consistent with a continuous medium. This dialectic coexistence of complexity and simplicity, discreetness and continuity suggests the existence of certain rule-based assignment, which 'may be applied equally well to all the ventricular myocardial fibers', enabling the ventricular myocardial mass to assemble abundant, dynamic, stochastic vectorial forces and produce apparently smooth, averaged, continuous, global response.

ELIGIBILITY:
Inclusion Criteria:

* Structurally normal mitral and aortic valve;
* Technically adequate color flow Doppler image;
* Technically adequate real-time 3D echocardiographic image of the LV chamber and the mitral apparatus (annulus and leaflets) to allow analysis of 3D geometry;
* Normal sinus rhythm.

Exclusion Criteria:

* Recurrent MI or coronary reintervention during the follow up period;
* Clinical or echocardiographic evidence of other cardiac diseases, such as organic valvular, pericardial, congenital, or infiltrative heart disease;
* Right ventricular alterations resulting in abnormal position or movement of the septum.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after AMI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-10; Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-chun Lin, Ph D, Study Director — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan